CLINICAL TRIAL: NCT02229175
Title: Comparison of Subvisible Retinal Laser Therapy With Intravitreal Bevacizumab in Treatment of Diabetic Macular Edema
Brief Title: Laser vs Bevacizumab Injection Alone in Treatment of Diabetic Macular Edema
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study not feasible with current resources.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-14153
Record Dates: First submitted 2014-08-14; First posted 2014-09-01 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; Diabetic Retinopathy; Type 1 Diabetes; Type 2 Diabetes; Macular Edema; bevacizumab; intravitreal injection; Avastin; PASCAL Endpoint Management (EpM) system; Subthreshold focal laser treatments
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Macular Edema | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IVB + laser (Experimental): Intravitreal bevacizumab (IVB) will be administered at baseline, month 1, and month 2, consistent with previous DME trials. Subvisible laser treatment will be administered at baseline. Patients will then undergo monthly surveillance, as they would with standard of care treatment, allowing for retreatment with monthly IVB and laser therapy every 3 months if defined retreatment criteria are met, as described below.
  Interventions: Drug: bevacizumab; Device: PASCAL Endpoint Management (EpM) laser treatment
- IVB only (Active Comparator): IVB monthly at baseline, month 1, and month 2. Patients will then undergo monthly surveillance, as they would with standard of care treatment, allowing for retreatment with monthly IVB if defined retreatment criteria are met, as described below. Patients will also undergo sham laser treatment (patient will be placed in front of laser but no laser will be activated) to mask the patient to the treatment.
  Interventions: Drug: bevacizumab

INTERVENTIONS:
Drug: bevacizumab — intravitreal injections of antibodies inhibiting vascular endothelial growth factor
  Other Names: Avastin
Device: PASCAL Endpoint Management (EpM) laser treatment — This is an algorithm that is included in the PASCAL 577 mm yellow laser system (Topcon, Santa Clara, CA). This is FDA-approved for treatment of diabetic retinopathy and diabetic macular edema.
  Arms: IVB + laser

SUMMARY:
Currently, diabetic macular edema is treated is through injection of a medications such as off-label bevacizumab, which decreases the swelling in the retina. These injections are sometimes required monthly until the condition is controlled. Recently, there have been some new FDA approved treatments using laser that decrease the swelling. These approximately ten minute treatments do not require injections and don't cause permanent damage to the eye, and they may decrease the number of injections one needs to get to treat diabetic macular edema (DME).

The purpose of this randomized clinical trial is to determine whether subvisible laser in combination with intravitreal bevacizumab is non-inferior compared to current standard of care (intravitreal bevacizumab alone) in achieving favorable outcomes for visual acuity, mean macular thickness, and patient quality of life, and has fewer needed intravitreal bevacizumab injections throughout the course of the 12 month study period.

DETAILED DESCRIPTION:
The patient is randomized into one of two study groups described below.

* Group 1: Intravitreal bevacizumab (IVB) will be administered at the first 3 monthly visits and subvisible laser treatment will be administered at the first visit. The the patient will undergo monthly visits, as he/she would with standard of care treatment, allowing for retreatment with monthly IVB and laser treatment every 3 months if defined retreatment criteria are met, as determined by a physician.
* Group 2: Intravitreal bevacizumab (IVB) will be administered at the first 3 monthly visits. The patient will then undergo monthly exams, as he or she would with standard of care treatment, allowing for retreatment with monthly IVB if defined retreatment criteria are met, as determined by a physician. The patient may also undergo sham laser treatment (he/she will be placed in front of laser but no laser will be activated) so that the patient isn't made aware of which treatment group he/she is a part of.

Other data that will be collected throughout the study at monthly examinations:

* Monthly Snellen Visual acuity test
* Monthly spectral-domain optical coherence tomography (SD-OCT) imaging using standard clinic protocol monthly
* Standard clinic diabetic montage Fundus photos at months 0,6,12
* Fluorescein angiography at months 0, 6, 12

The subjects' visit schedules will be the same as for routine standard of care for the IVB injection procedure. There are no additional appointments for this study.

All study procedures will be done at San Francisco General Hospital

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include adults ≥ 18 years with type 1 or 2 diabetes mellitus with DME secondary to diabetes mellitus involving the center of the macula in the study eye and with a decrease in vision is determined to be primarily the result of DME in the study eye. The study eye must have a BCVA ETDRS letter score of 50 to 24 (20/30 to 20/320) in the study eye. The patient should be on a stable medical diabetic regimen that is not expected to change.

Exclusion Criteria:

* Patients are excluded if they have had laser photocoagulation (panretinal or macular) in the study eye within 90 days of Day 1, more than two previous macular laser treatments in the study eye, previous use of intraocular or periocular corticosteroids in the study eye within 90 days of Day 1, previous treatment with antiangiogenic drugs in either eye (pegaptanib sodium, bevacizumab, ranibizumab, or aflibercept) within 45 days of Day 1, active proliferative diabetic retinopathy (PDR) in the study eye, with the exception of inactive, regressed PDR, uncontrolled diabetes mellitus, as defined by HbA1c > 12%, or a patient who is functionally monocular, as defined by the clinician or vision worse than 20/400 in the fellow eye even if that eye is otherwise eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Retinal thickness | 12 months
  Change in retinal thickness on SD-OCT from baseline to 12 months.

SECONDARY OUTCOMES:
Visual Acuity | 12 months
  Change in Snellen visual acuity from baseline to 12 months.
Number of injections of bevacizumab needed | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jay Stewart, MD, Principal Investigator — University of California, San Francisco; Daniel Chao, MD, PhD, Principal Investigator — University of California, San Diego; Catherine Psaras, BA, Study Director — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States